CLINICAL TRIAL: NCT01567345
Title: Comparison of Two Types of Intrathecal Morphine Administration by Pump for Analgesia in Cancer Patients With Failure of Conventional Analgesic Therapy.
Brief Title: Intrathecal Morphine Administration Using Implantable Pump With Continuous or Programmable Flow
Acronym: PITAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPP-401; 2008-005087-14 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-03-30 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Advanced Cancer; Intractable Pain
Keywords: Pain; cancer; Intrathecal; analgesia; Morphine; Implantable pump
MeSH Terms: conditions — Pain, Intractable; Pain; Neoplasms; Agnosia | interventions — Infusion Pumps, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal pump with continuous flow (Active Comparator): After placement of the implantable pump, continuous flow is scheduled by physician and the patient can't modify it.
  Interventions: Device: Implantable pump with continuous flow
- Intrathecal pump with programmable flow. (Experimental): After placement of the implantable pump, programmable flow is scheduled by physician and patient can do himself morphine bolus injections for a better control of acute episodes of pain.
  Interventions: Device: Implantable pump with programmable flow.

INTERVENTIONS:
Device: Implantable pump with continuous flow — Insertion of an implantable pump filled up with the analgesic solution. Connection of the catheter to the intrathecal space. Continuous morphine's flow is scheduled.
  Other Names: Isomed Pump 8472
  Arms: Intrathecal pump with continuous flow
Device: Implantable pump with programmable flow. — Insertion of an implantable pump filled up with the analgesic solution. Connection of the catheter to the intrathecal space. Programmable morphine's flow is scheduled.
  Other Names: Synchromed II pump 8637
  Arms: Intrathecal pump with programmable flow.

SUMMARY:
The aim of this study is to compare intrathecal morphine administration: using a pump with continuous or programmable flow.

DETAILED DESCRIPTION:
Cancer is frequently associated with pain. In spite of recent improvements in cancer related pain treatment, incidence of cancerous chronic pain did not decrease. Indeed, 15 to 20% of patients are still suffering from intractable pain despite an optimal symptom management.

Treatment of cancer pain is generally based on the WHO analgesic ladder according to 3 steps. Patients with advanced cancer are often treated at WHO step 3 analgesics, i.e. morphine and its derivatives, at high dosages. But increasing the dosage of opioids also leads to accentuation of their adverse events and the corresponding risks.

At this stage of the disease, in patients with failure of conventional analgesic therapy, intrathecal injection of analgesics can be decided in order to relieve pain. 2 types of pumps allow intrathecal morphine administration : continuous or programmable flow. In this study, we want to compare the quality of analgesia obtained through these 2 flows.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old.
* Patient with advanced cancer.
* Patient with severe pain, i.e. a mean daily pain score > or = 5 on an numeric rating scale.
* Failure of optimal conventional analgesic therapy : either due to intolerable adverse events or to lack of efficacy, i.e. after having tried opioid rotation techniques, different way of administration, use of rapid-acting narcotics to control acute episodes of pain, use of intravenous morphine by PCA pump.
* Possibility of return home
* Dated and signed informed consent form.

Exclusion Criteria:

* Patient's refusal to participate in the study.
* Ongoing pregnancy.
* Ongoing systemic infection.
* Injection site infection.
* Estimated survival less than 90 days.
* Allergy or intolerance to morphine.
* Contraindication to implantation of an intrathecal catheter.
* Patient treated with a powerful CYP1A2 inhibitor, such as fluvoxamine or enoxacin.
* Intrathecal chemotherapy planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-01-14 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pain improvement between 2 groups. | At 3 month
  Pain will be assessed every day by patient using a Visual Analog Scale (VAS. VAS scores will be compared between 2 groups(continuous or programmable flow). We want to demonstrate the superiority of intrathecal analgesia obtained through programmable flow compared to continuous flow.

SECONDARY OUTCOMES:
Pain improvement with intrathecal analgesia compared to previous antalgic therapy. | at 3 month
  Using Visual Analog Scale's score, we want to demonstrate the superiority of intrathecal analgesia compared to previous treatment (pain is assessed through VAS within 4 days before inclusion).
Adverse Events assessment. | every month
  We want to demonstrate a reduction of adverse events related to intrathecal analgesia compared to the previous treatment and to compare the two delivery systems.
  Adverse events due to morphine (6 types) will be scored according to 4 levels, then the sum of these scores will constitute an adverse event severity index ranging from 0 to 18. This index will be compared between the 2 arms and will also be compared to baseline values before introduction of intrathecal analgesia.
Patient's performance status improvement. | At 1 month
  We want to demonstrate improvement of the patient's performance status during intrathecal analgesia compared to the previous treatment and to compare the two delivery systems.
Incidence and types of complications. | every month.
  We want to compare the incidence and type of complications (infectious, morphine-related and co-analgesic treatments-related, due to the intrathecal catheter, to the implantable pump) between the two delivery systems.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Dupoiron, MD, Principal Investigator — Institut Cancerologie de l'Ouest
Locations (6):
- France (6):
  - ICO Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier, Laon
  - Centre Oscar Lambret, Lille
  - Hôpital Laennec, Nantes
  - Polyclinique, Poitiers